CLINICAL TRIAL: NCT00581100
Title: Randomised, Open-label Preliminary Study to Assess the Effects of 2 Regimens of Etanercept on Nail and Skin Symptoms in Patients With Nail Psoriasis and Plaque Psoriasis
Brief Title: Effects of Etanercept on Nail Psoriasis and Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0881A6-409
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Results first posted 2010-08-30 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Nail Psoriasis; Plaque Psoriasis
Keywords: Nail Psoriasis; Plaque Psoriasis
MeSH Terms: interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): etanercept 50 mg SC injection twice weekly for 12 weeks reducing to etanercept 50 mg once weekly to week 24
  Interventions: Drug: etanercept
- 2 (Active Comparator): etanercept 50 mg SC once weekly for the complete 24 week treatment period
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept — Subjects randomized to Arm 1 shall be treated with ETN 50 mg twice weekly for 12 weeks reducing thereafter to ETN 50 mg once weekly to 24 weeks.
  Subjects randomized to Arm 2 shall be treated with ETN 50 mg once weekly for the entire 24 week treatment period.

SUMMARY:
The purpose of this study is to evaluate if Etanercept administered at a higher initial dose provides greater improvement in nail and skin psoriasis symptoms than a regimen with a lower initial dose.

DETAILED DESCRIPTION:
This study will assess the effects of the 2 Etanercept regimens on fingernail psoriasis over 24 weeks among patients with both skin and fingernail symptoms who have previously failed at least one therapy for nail psoriasis. The endpoint of 24 weeks was chosen to allow sufficient time for normal nail growth.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Active, stable plaque psoriasis defined by the following criteria:

  * Body surface area (BSA) ≥ 10 % at screening and baseline
  * Or, PASI >10 at screening and baseline
  * Or, PGA of Psoriasis status of moderate or worse (moderate, marked, or severe) at screening and baseline
  * Or, DLQI > 10 at baseline
* Active fingernail psoriasis defined as target fingernail NAPSI ≥ 2 and overall NAPSI > 14 - Target nail is defined as the nail with the highest nail score (matrix+bed scores) at baseline. Should more than one fingernail have the same score, the target fingernail will be chosen by the investigator.
* Failure of at least one systemic psoriasis therapy for nail psoriasis
* Eligible to receive biologic therapy for psoriasis in accordance to local guidelines

Exclusion Criteria:

* Evidence of Skin conditions other than psoriasis
* Psoralen plus ultraviolet radiation (PUVA), cyclosporine, alefacept, methotrexate, acitretin, or any other systemic anti-psoriasis therapy within 28 days of study drug initiation
* Prior exposure to any TNF-inhibitor. Prior exposure to efalizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2007-09; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eighty-five participants were screened for the study; 13 participants were screening failures, and 72 participants were randomized to treatment.
Groups:
- Etanercept: Twice, Then Once Weekly: Etanercept 50 mg subcutaneous (SC) injection twice weekly for 12 weeks reduced to Etanercept 50 mg once weekly to week 24
- Etanercept: Once Weekly: Etanercept 50 mg SC once weekly for the complete 24 week treatment period
Period: Overall Study
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly
Started | 38 | 34
Modified Intent-To-Treat Population | 36 (At least one dose of study medication, and had baseline and post-baseline data.) | 33 (At least one dose of study medication, and had baseline and post-baseline data.)
Completed | 31 | 29
Not Completed | 7 | 5
Not completed — Death | 1 | 0
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Other | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly | Total
Number analyzed (Participants) | 36 | 33 | 69
Age, Customized [Mean (Standard Deviation); unit: years] | 46.28 (13.51) | 45.36 (9.19) | 45.84 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 26 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Nail Psoriasis Severity Index (NAPSI) Score for Target Fingernail
Description: Target fingernail (highest matrix + bed scores at baseline) divided with imaginary lines into quadrants and graded for nail matrix and nail bed psoriasis. Sum of scores = total score for that nail (0-8). Nail Matrix Psoriasis = pitting, leukonychia, red spots in lunula, and/or nail plate crumbling. Nail Bed Psoriasis = onycholysis, splinter hemorrhages, oil drop (salmon patch) discoloration, and/or nail bed hyperkeratosis. Range for both scores: 0 (none), 1 (present in 1/4 nail), 2 (present in 2/4 nail), 3 (present in 3/4 nail), 4 (present in 4/4 nail). Higher scores = more severe psoriasis.
Time Frame: Baseline, Week 24
Population: Modified Intent-to-Treat (mITT) population: all randomized participants who received at least one dose of study medication, and provided baseline and post-baseline data. N = number of participants with evaluable data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly
Number analyzed (Participants) | 35 | 32
units on a scale | -4.32 [-4.91 to -3.73] | -4.36 [-4.98 to -3.74]
Statistical Analysis 1: Comparison: Etanercept: Twice, Then Once Weekly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted change calculated from mixed-model. Model for change = [Group visit Group*visit baseline baseline*visit]
Statistical Analysis 2: Comparison: Etanercept: Once Weekly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Adjusted change calculated from mixed-model. Model for change = [Group visit Group*visit baseline baseline*visit]

2. Secondary Outcome: Change From Baseline in Overall Nail Psoriasis Severity Index (NAPSI) Score
Description: NAPSI (matrix + bed score) performed on dorsal views of 8 fingers, excluding thumb; range: 0 to 8. Overall NAPSI score = sum of all fingernail scores; range: 0 to 64. Nails were divided into quadrants and graded for nail matrix and bed psoriasis. Nail Matrix Psoriasis = pitting, leukonychia, red spots in lunula, and/or nail plate crumbling. Nail Bed Psoriasis = onycholysis, splinter hemorrhages, oil drop (salmon patch) discoloration, and/or nail bed hyperkeratosis. Range for both scores: 0 (none), 1 (present 1/4 nail), 2 (present 2/4 nail), 3 (present 3/4 nail), and 4 (present 4/4 nail).
Time Frame: Baseline, Week 24
Population: mITT, N = number of participants with evaluable data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly
Number analyzed (Participants) | 35 | 32
units on a scale | -22.64 [-26.44 to -18.85] | -22.63 [-26.61 to -18.66]
Statistical Analysis 1: Comparison: Etanercept: Twice, Then Once Weekly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted change calculated from mixed-model. Model for change = [Group visit Group*visit baseline baseline*visit]
Statistical Analysis 2: Comparison: Etanercept: Once Weekly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Adjusted change calculated from mixed-model. Model for change = [Group visit Group*visit baseline baseline*visit]

3. Secondary Outcome: Percent of Participants Who Achieved a 50% Improvement in the Nail Psoriasis Severity Index (NAPSI) Score for Target Fingernail at Week 12 and Week 24
Description: Target fingernail (highest matrix + bed scores at baseline) divided with imaginary lines into quadrants and graded for nail matrix and nail bed psoriasis. Sum of scores = total score for that nail (0-8). Nail Matrix Psoriasis = pitting, leukonychia, red spots in lunula, and/or nail plate crumbling. Nail Bed Psoriasis = onycholysis, splinter hemorrhages, oil drop (salmon patch) discoloration, and/or nail bed hyperkeratosis. Range for both scores 0-8: 0 (none), 1 (present in 1/4 nail), 2 (present in 2/4 nail), 3 (present in 3/4 nail),4 (present in 4/4 nail). Higher score = more severe psoriasis.
Time Frame: Week 12, Week 24
Population: mITT, N = number of participants with evaluable data.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly
Number analyzed (Participants) | 36 | 33
percent of participants
  Week 12 | 60.61 | 51.61
  Week 24 | 82.86 | 81.25
Statistical Analysis 1: Comparison: Etanercept: Twice, Then Once Weekly; Week 12; Test type: Superiority or Other; p < 0.001, GEE model — P-value from generalized linear models for correlated data using Generalized Estimating Equations (GEE), with treatment and visits as fixed factors. Model for proportion = [Group visit Group*visit]
Statistical Analysis 2: Comparison: Etanercept: Once Weekly; Week 12; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Etanercept: Twice, Then Once Weekly; Week 24; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Etanercept: Once Weekly; Week 24; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 3, analysis 1]

4. Secondary Outcome: Percent of Participants Who Achieved a 75% Improvement in the Nail Psoriasis Severity Index (NAPSI) Score for Target Fingernail at Week 12 and Week 24
Description: as for outcome 1
Time Frame: Week 12, Week 24
Population: mITT, N = number of participants with evaluable data.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly
Number analyzed (Participants) | 36 | 33
percent of participants
  Week 12 | 18.18 | 19.35
  Week 24 | 57.14 | 68.75
Statistical Analysis 1: Comparison: Etanercept: Twice, Then Once Weekly; Week 12; Test type: Superiority or Other; p = 0.007, GEE model — P-value from generalized linear models for correlated data using Generalized Estimating Equations (GEE) with treatment and visits as fixed factors. Model for proportion=[Group visit Group*visit]
Statistical Analysis 2: Comparison: Etanercept: Once Weekly; Week 12; Test type: Superiority or Other; p = 0.006, GEE model — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Etanercept: Twice, Then Once Weekly; Week 24; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Etanercept: Once Weekly; Week 24; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 4, analysis 1]

5. Secondary Outcome: Percent of Participants Who Achieved a 50% Improvement in the Nail Psoriasis Severity Index (NAPSI) for Overall NAPSI Score at Week 12 and Week 24
Description: as for outcome 2
Time Frame: Week 12, Week 24
Population: mITT, N = number of participants with evaluable data.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly
Number analyzed (Participants) | 36 | 33
percent of participants
  Week 12 | 54.55 | 48.39
  Week 24 | 68.57 | 81.25
Statistical Analysis 1: Comparison: Etanercept: Twice, Then Once Weekly; Week 12; Test type: Superiority or Other; p < 0.001, GEE model — P-value from generalized linear models for correlated data using Generalized Estimating Equations (GEE), with treatment and visits as fixed factors. Model for proportion =[Group visit Group*visit]
Statistical Analysis 2: Comparison: Etanercept: Once Weekly; Week 12; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Etanercept: Twice, Then Once Weekly; Week 24; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Etanercept: Once Weekly; Week 24; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 5, analysis 1]

6. Secondary Outcome: Percent of Participants Who Achieved a 75% Improvement in the Nail Psoriasis Severity Index (NAPSI) for Overall NAPSI Score at Week 12 and Week 24
Description: as for outcome 2
Time Frame: Week 12, Week 24
Population: mITT, N = number of participants with evaluable data.
Measure: Number; unit: units on a scale
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly
Number analyzed (Participants) | 36 | 33
units on a scale
  Week 12 | 9.09 | 19.35
  Week 24 | 62.86 | 62.50
Statistical Analysis 1: Comparison: Etanercept: Twice, Then Once Weekly; Week 12; Test type: Superiority or Other; p = 0.069, GEE model — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Etanercept: Once Weekly; Week 12; Test type: Superiority or Other; p = 0.006, GEE model — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Etanercept: Twice, Then Once Weekly; Week 24; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Etanercept: Once Weekly; Week 24; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 4, analysis 1]

7. Secondary Outcome: Change From Baseline in the Psoriasis Area and Severity Index (PASI) Score
Description: Combined assessment of lesion severity and area affected into single score; range: 0 (no disease) to 72 (maximal disease). Body was divided into 4 sections (head, arms, trunk, legs); each area was scored by itself and scores were combined for final PASI. For each section percent (%) area of skin involved was estimated: 0 (0%) to 6 (90 - 100%), and severity was estimated by clinical signs: erythema, induration, and desquamation; scale: 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each section * area score * weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4).
Time Frame: Baseline, Week 24
Population: mITT, N = number of participants with evaluable data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly
Number analyzed (Participants) | 35 | 32
units on a scale | -14.81 [-16.56 to -13.05] | -14.11 [-15.95 to -12.28]
Statistical Analysis 1: Comparison: Etanercept: Twice, Then Once Weekly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Adjusted change calculated from mixed model. Model for change=[Group visit group*visit baseline baseline*visit]
Statistical Analysis 2: Comparison: Etanercept: Once Weekly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Adjusted change calculated from mixed model. Model for change=[Group visit group*visit baseline baseline*visit]

8. Secondary Outcome: Percent of Participants Achieving a 50% Improvement in the Psoriasis Area and Severity Index (PASI) Score at Week 12 and Week 24
Description: as for outcome 7
Time Frame: Week 12 , Week 24
Population: mITT, N = number of participants with evaluable data.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly
Number analyzed (Participants) | 36 | 33
percent of participants
  Week 12 | 90.91 | 87.10
  Week 24 | 85.71 | 84.38
Statistical Analysis 1: Comparison: Etanercept: Twice, Then Once Weekly; Week 12; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Etanercept: Once Weekly; Week 12; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Etanercept: Twice, Then Once Weekly; Week 24; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Etanercept: Once Weekly; Week 24; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 4, analysis 1]

9. Secondary Outcome: Percent of Participants Achieving a 75% Improvement in the Psoriasis Area and Severity Index (PASI) Score at Week 12 and Week 24
Description: as for outcome 7
Time Frame: Week 12 , Week 24
Population: mITT, N = number of participants with evaluable data.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly
Number analyzed (Participants) | 36 | 33
percent of participants
  Week 12 | 51.52 | 58.06
  Week 24 | 77.14 | 62.50
Statistical Analysis 1: Comparison: Etanercept: Twice, Then Once Weekly; Week 12; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Etanercept: Once Weekly; Week 12; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Etanercept: Twice, Then Once Weekly; Week 24; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Etanercept: Once Weekly; Week 24; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 4, analysis 1]

10. Secondary Outcome: Change From Baseline in Physician Global Assessment (PGA) of Psoriasis
Description: Physician Global Assessment (PGA) of Psoriasis: score based on dermatologist's assessment of disease averaged over all lesions of head, scalp, and neck. Overall lesions were graded for induration, erythema, and scaling; range: 0 (no evidence) to 5 (severe). The sum of the 3 scores was divided by 3 to obtain a final PGA score. Higher scores indicate greater severity of disease.
Time Frame: Baseline, Week 24
Population: mITT, N = number of participants with evaluable data.
Measure: Mean (95% Confidence Interval); unit: unts on a scale
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly
Number analyzed (Participants) | 35 | 32
unts on a scale | -1.65 [-2.05 to -1.26] | -1.84 [-2.25 to -1.43]
Statistical Analysis 1: Comparison: Etanercept: Twice, Then Once Weekly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Adjusted change calculated from mixed model. Model for change-[Group visit Group*visit baseline baseline*visit]
Statistical Analysis 2: Comparison: Etanercept: Once Weekly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Adjusted change calculated from mixed model. Model for change-[Group visit Group*visit baseline baseline*visit]

11. Secondary Outcome: Percent of Participants Achieving a Status on the Physician Global Assessment (PGA) of Psoriasis of Clear or Almost Clear
Description: Physician Global Assessment (PGA) of Psoriasis: score based on dermatologist's assessment of disease averaged over all lesions of head, scalp, and neck. Overall lesions were graded for induration, erythema, and scaling; range: 0 (no evidence) to 5 (severe). The sum of the 3 scores was divided by 3 to obtain a final PGA score. Higher scores indicate greater severity of disease. Assessment of clear or almost clear = PGA score of 0 (no evidence), or 1 (minimal/faint).
Time Frame: Baseline, Week 24 or Early Termination
Population: mITT, N = number of participants with evaluable data.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly
Number analyzed (Participants) | 35 | 32
percent of participants | 68.57 | 75.00
Statistical Analysis 1: Comparison: Etanercept: Twice, Then Once Weekly; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Etanercept: Once Weekly; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 4, analysis 1]

12. Secondary Outcome: Percent of Participants Achieving a Status on the Physician Global Assessment (PGA) of Psoriasis of Mild or Better
Description: Physician Global Assessment (PGA) of Psoriasis: score based on dermatologist's assessment of disease averaged over all lesions of head, scalp, and neck. Overall lesions were graded for induration, erythema, and scaling; range: 0 (no evidence) to 5 (severe). The sum of the 3 scores was divided by 3 to obtain a final PGA score. Higher scores indicate greater severity of disease. Assessment of mild or better = PGA score of ≤ 2 (mild plaque elevation, mild scaling, and light red coloration).
Time Frame: Baseline, Week 24 or Early Termination
Population: mITT, N = number of participants with evaluable data.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly
Number analyzed (Participants) | 35 | 32
percent of participants | 82.86 | 87.50
Statistical Analysis 1: Comparison: Etanercept: Twice, Then Once Weekly; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Etanercept: Once Weekly; Test type: Superiority or Other; p < 0.001, GEE model — [p-value comment as in outcome 4, analysis 1]

13. Secondary Outcome: Change From Baseline in the Dermatology Life Quality Index (DLQI)
Description: Self-administered questionnaire to measure health-related quality of life (QoL)of adult patients suffering from skin disease; 10 questions concerning patients' perception of impact of their disease over last week encompassing aspects such as symptoms, feelings, daily activities, leisure, work, school, personal relationships and side effects of treatment. Questions scored on a 4-point Likert scale: 0 (not at all/not relevant), 1 (a little), 2 (a lot), and 3 (very much). Scores of individual items (0-3) were added to yield a total score (0-30); higher score = greater impairment of patient's QoL.
Time Frame: Baseline, Week 24
Population: mITT, N = number of participants with evaluable data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly
Number analyzed (Participants) | 35 | 31
units on a scale | -8.60 [-9.98 to -7.21] | -8.74 [-10.21 to -7.26]
Statistical Analysis 1: Comparison: Etanercept: Twice, Then Once Weekly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Adjusted change calculated from mixed-model. Model for change=[Group visit Group*visit baseline baseline*visit]
Statistical Analysis 2: Comparison: Etanercept: Once Weekly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Adjusted change calculated from mixed-model. Model for change=[Group visit Group*visit baseline baseline*visit]

14. Secondary Outcome: Change From Baseline in Physician Assessment of Nail Psoriasis Activity Visual Analog Scale (VAS)
Description: Physician global assessment of disease activity using a visual analog scale; range: 0 (no nail disease) to 100 (worst possible nail disease).
Time Frame: Baseline, Week 24
Population: mITT, N = number of participants with evaluable data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly
Number analyzed (Participants) | 34 | 32
units on a scale | -44.66 [-52.11 to -37.21] | -41.03 [-48.70 to -33.35]
Statistical Analysis 1: Comparison: Etanercept: Twice, Then Once Weekly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Adjusted change calculated from mixed model. Model for change=[Group visit Group*visit baseline baseline*visit]
Statistical Analysis 2: Comparison: Etanercept: Once Weekly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Adjusted change calculated from mixed model. Model for change=[Group visit Group*visit baseline baseline*visit]

15. Secondary Outcome: Change From Baseline in Patient Assessment of Nail Psoriasis Activity Visual Analog Scale (VAS)
Description: Patient global assessment of disease activity using a visual analog scale; range: 0 (no nail disease) to 100 (worst possible nail disease).
Time Frame: Baseline, Week 24
Population: mITT, N = number of participants with evaluable data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly
Number analyzed (Participants) | 35 | 32
units on a scale | -48.89 [-56.86 to -40.91] | -41.69 [-50.02 to -33.35]
Statistical Analysis 1: Comparison: Etanercept: Twice, Then Once Weekly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Adjusted change calculated from mixed model. Model for change=[Group visit Group*visit baseline baseline*visit]
Statistical Analysis 2: Comparison: Etanercept: Once Weekly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — <Table 8-14> Change from baseline in Physician and Patient Assessment of Nail Psoriasis Activity Visual Analog Scale (VAS)

16. Secondary Outcome: Change From Baseline in Physician Fingernail Grading Assessment Total Score
Description: Physician assessment of disease activity for each fingernail; range: 0 (no disease), 1 (mild disease, 2 (moderate disease), or 3 (severe disease). Total score range = 0-30.
Time Frame: Baseline, Week 24
Population: mITT, N = number of participants with evaluable data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly
Number analyzed (Participants) | 35 | 32
units on a scale | -11.47 [-13.54 to -9.41] | -12.21 [-14.37 to -10.05]
Statistical Analysis 1: Comparison: Etanercept: Twice, Then Once Weekly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Adjusted change calculated from mixed-model. Model for change=[Group visit Group*visit baseline baseline*visit]
Statistical Analysis 2: Comparison: Etanercept: Once Weekly; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Adjusted change calculated from mixed-model. Model for change=[Group visit Group*visit baseline baseline*visit]

ADVERSE EVENTS:
Description: Safety population: all subjects who took at least one dose of study medication.
Arm/Group | Etanercept: Twice, Then Once Weekly | Etanercept: Once Weekly
Serious Adverse Events (participants affected / at risk) | 2/38 | 0/34
Other Adverse Events (participants affected / at risk) | 22/38 | 12/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept: Twice, Then Once Weekly (N=38) | Etanercept: Once Weekly (N=34)
Lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept: Twice, Then Once Weekly (N=38) | Etanercept: Once Weekly (N=34)
Leukocytosis not otherwise specified (NOS) (Blood and lymphatic system disorders) | 1 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0
Conjunctivitis NEC (Eye disorders) | 0 | 1
Hyperacidity (Gastrointestinal disorders) | 1 | 0
Abdominal pain NOS (Gastrointestinal disorders) | 1 | 0
Vomiting NOS (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea NOS (Gastrointestinal disorders) | 1 | 0
Loose stools (Gastrointestinal disorders) | 0 | 1
Sore throat NOS (Gastrointestinal disorders) | 1 | 0
Injection site dermatitis (General disorders) | 1 | 1
Injection site pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 2 | 1
Application site rash (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Injection site burning (General disorders) | 1 | 0
Injection site urticaria (General disorders) | 1 | 0
Liver fatty (Hepatobiliary disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 4
Tooth abscess (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1
Respiratory tract infection NOS (Infections and infestations) | 1 | 0
Pharyngitis NOS (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 1
Transaminase NOS increased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Localized osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Localized infection (Infections and infestations) | 1 | 0
Headache NOS (Nervous system disorders) | 4 | 3
Burning sensation NOS (Nervous system disorders) | 0 | 1
Paraesthesia NEC (Nervous system disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus NOS (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis aggravated (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder NOS (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hematoma NOS (Vascular disorders) | 1 | 0
Hypertension NOS (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.